CLINICAL TRIAL: NCT07042997
Title: Evaluation of Anatomical Accuracy in Targeting Forearm Extensor Muscles With Blind Dry Needling in Patients With Lateral Epicondylitis Using Ultrasound Guidance
Brief Title: Ultrasound Evaluation of Blind Dry Needling in Lateral Epicondylitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: nurmuhammet tas (Other Government)
Responsible Party: Sponsor-Investigator, nurmuhammet tas, DR., Erzurum Regional Training & Research Hospital
Organization: Erzurum Regional Training & Research Hospital (Other Government)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ErzurumNMT
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Lateral Epicondylitis
Keywords: lateral epicondylitis; dry needling; trigger point; ultrasound guidance
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- lateral epicondylitis and with at least one active trigger point (Experimental): The first clinician determines the active TrP by manual palpation and performs dry needling without the use of ultrasound (blinded).
  Interventions: Procedure: Evaluation of Anatomical Accuracy in Targeting Forearm Extensor Muscles with Blind Dry Needling in Patients with Lateral Epicondylitis Using Ultrasound Guidance
- Ultrasound-Guided Needle Location Verification (Experimental): After the needling procedure, a second clinician evaluates the needle's location in the muscle using ultrasonography.
  Interventions: Procedure: Evaluation of Anatomical Accuracy in Targeting Forearm Extensor Muscles with Blind Dry Needling in Patients with Lateral Epicondylitis Using Ultrasound Guidance

INTERVENTIONS:
Procedure: Evaluation of Anatomical Accuracy in Targeting Forearm Extensor Muscles with Blind Dry Needling in Patients with Lateral Epicondylitis Using Ultrasound Guidance — Using a high-resolution linear probe (5-12 MHz) , the muscle in which the needle tip is located is monitored in real time in the transverse and longitudinal planes. Whether the needle is in the targeted muscle is recorded as "correct" or "incorrect".

SUMMARY:
The aim of this clinical study is to evaluate the accuracy and consistency of the blinded needling procedure by evaluating the dry needling procedure under ultrasound guidance in patients diagnosed with lateral epicondylitis and with at least one active trigger point (MTrP) in the forearm extensor muscles. The study is a prospective, double-blind validation study.

Participants: Volunteers aged 18-70 years, who have pain in the lateral epicondyle region for at least 6 weeks and who have active trigger points in the forearm extensor muscles detected by physical examination will be included in the study. Written informed consent will be obtained from all participants.

DETAILED DESCRIPTION:
Muscle Selection and Application Protocol All patients will be prescribed nonsteroidal anti-inflammatory (NSAID) and analgesic treatments in accordance with clinical standards, and the use of a wrist splint will be recommended to support symptom control. Four muscles are targeted during the evaluation: Extensor carpi radialis brevis (ECRB), Extensor carpi radialis longus (ECRL), Extensor digitorum communis (EDC), and Brachioradialis (BR).

Blinded Dry Needling Application The first clinician determines the active TrP by manual palpation and performs dry needling without the use of ultrasound (blinded). The needling procedure is performed in accordance with the intramuscular TrP localization and techniques in Myofascial Pain and Dysfunction: The Trigger Point Manual.

The patient is placed in the supine position. The needle used is a Hua - Long brand 0.30 x 30 mm single-use sterile acupuncture needle. The needle is advanced to the TrP and modulated until a local twitch response is obtained. If the patient experiences significant discomfort, the procedure is terminated.

Ultrasound-Guided Needle Location Verification After the needling procedure, a second clinician evaluates the needle's location in the muscle using ultrasonography. This clinician is blinded to the target muscle. Imaging is performed in accordance with the guidance of 'Ultrasound of the Musculoskeletal System' Using a high-resolution linear probe (5-12 MHz) , the muscle in which the needle tip is located is monitored in real time in the transverse and longitudinal planes. Whether the needle is in the targeted muscle is recorded as "correct" or "incorrect".

ELIGIBILITY:
Inclusion Criteria:

* Volunteers aged 18-70 years,
* who have pain in the lateral epicondyle region for at least 6 weeks
* who have active trigger points in the forearm extensor muscles detected by physical examination

Exclusion Criteria:

* Those who have not complained of pain in the lateral epicondyle region for at least 6 weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-21 (Estimated); Primary Completion 2025-09-22 (Estimated); Study Completion 2025-09-23 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Anatomical Accuracy in Targeting Forearm Extensor Muscles with Blind Dry Needling in Patients with Lateral Epicondylitis Using Ultrasound Guidance | 2 week
  Correct placement rates will be calculated for each muscle. The agreement between the ultrasound and verification results of the blinded applications will be evaluated with Kappa statistics. Chi-square test or McNemar test will be used for differences between muscles.